CLINICAL TRIAL: NCT04610814
Title: Blood Transfusion by Boston MedFlight Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston MedFlight (Unknown); Boston Medical Center (Other); Tufts Medical Center (Other); Lahey Clinic (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Susan Renee Wilcox, Chief, Division of Critical Care, Department of Emergency Medicine, Massachusetts General Hospital
Other Study IDs: 2019P003733
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Hemorrhagic Shock
Keywords: Blood transfusion; Pre-hospital care
MeSH Terms: conditions — Shock, Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Blood products during transport: Administration of appropriate blood products during transport
- Standard of Care: Receiving standard prehospital air medical care

SUMMARY:
The primary aim of this observational registry is to study the outcomes of patients with hemorrhagic shock transported by Boston MedFlight receiving blood products during transport.

DETAILED DESCRIPTION:
Boston MedFlight, a critical care transport organization, based on a consortium of the academic medical centers in Boston, will begin carrying PRBC in 2019. The program is intended to provide BMF clinicians with 24-hour immediate access to appropriate blood products to be utilized if needed for patients following life-threatening illness or injury. The four fundamental goals of this program are: save lives' ensure transfusion safety; minimize blood product waste; and conduct continuous quality assurance. Our goal is to observationally evaluate this new protocol of administering blood products in the pre-hospital setting. We will collect data on patients with hemorrhagic shock being transported by Boston MedFlight, who receive or would have been eligible to receive pre-hospital blood transfusion by the inclusion criteria.

ELIGIBILITY:
Inclusion criteria:

* Adult patients who would be eligible to receive blood products;

  * systolic blood pressure <90 mmHg
  * a shock index of > 0.9
  * clinical signs of shock as determined by the transport clinicians.

Exclusion Criteria:

* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient being transported by Boston MedFlight with hemorrhagic shock
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  30-day all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Susan R Wilcox, MD, Principal Investigator — Massachusetts General Hospital and Boston MedFlight
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States